CLINICAL TRIAL: NCT00827606
Title: A Three Year, Prospective, Open-label, Study To Evaluate Clinical Efficacy, Safety And Tolerability Of Atorvastatin In Children And Adolescents With Heterozygous Familial Hypercholesterolemia
Brief Title: Atorvastatin Three Year Pediatric Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2581173; 2008-006130-95 (EudraCT Number)
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Familial Hypercholesterolemia
Keywords: pediatric heterozygous familial hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atorvastatin (Experimental): All subjects will be treated with atorvastatin
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin tablets or chewable tablets, 5, 10, 20, 40 mg strengths, once daily, for three years (an 80 mg maximum daily dose is delivered by taking two 40 mg strengths, once daily)

SUMMARY:
The purpose of this study is to characterize three year descriptive growth and development (ie, height, weight, body mass index, Tanner Stage) and efficacy of cholesterol reduction in pediatric subjects with Heterozygous Familial Hypercholesterolemia receiving atorvastatin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Heterozygous familial hypercholesterolemia, ages 6-15, LDL greater than 4 mmol/l

Exclusion Criteria:

* Active liver disease or hepatic dysfunction, or persistent elevations of serum transaminases exceeding three times the upper limit of normal (ULN).

Female of childbearing potential who is not using adequate contraceptive measures or any female who is pregnant or breastfeeding. Any female who becomes pregnant during study participation will be immediately discontinued from treatment and counseled appropriately about the in utero exposure.

Known hypersensitivities to HMG-CoA reductase inhibitors

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 272 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (7):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - MEDPACE Clinical Pharmacology Unit, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Belgium (2):
  - Cliniques Universitaires Saint-Luc / Pediatrie generale, Brussels
  - Universitaire Ziekenhuizen Leuven / Center for Metabolic Diseases, Leuven
- Canada (2):
  - Clinique des Maladies Lipidiques de Quebec, Québec, Quebec
  - Clinique des maladies lipidiques de Quebec Inc, Sainte-Foy, Quebec
- Germany (2):
  - Charite Campus Virchow-Klinikum, Berlin
  - Augenaerztliche Gemeinschaftspraxis, Freiburg im Breisgau
- 1st Pediatrics Clinic , University of Athens, Agia Sofia Hospital, Athens, Greece
- Hungary (2):
  - Semmelweis Medical University, Budapest
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
- Italy (2):
  - Dipartimento di Medicina Clinica e delle Patologie Emergenti-University Hospital of Palermo, Palermo
  - Dipartimento di Clinica e Terapia Medica, Università degli Studi di Roma La Sapienza, Roma
- Rikshospitalet Lipidklinikken, Oslo, Norway
- Poland (2):
  - Poradnia Chorob Metabolicznych, Bydgoszcz
  - Klinika Chorob Metabolicznych, Warsaw
- Hospital de la Concepcion, San Germán, Puerto Rico
- Russia (4):
  - Moscow State Healthcare Institution 'Morozovskaya Children's City Clinical Hospital', Moscow
  - Autonomous Non-Profit Organization Medical Center 21 Century, Saint Petersburg
  - Saint-Petersburg State Pediatric Medical Academy, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution "Children's Polyclinic #35", Saint Petersburg
- Slovakia (5):
  - Metabolicka ambulancia, 2. Detská klinika Lekárskej fakulty Univerzity Komenského, Bratislava
  - Detska fakultna nemocnica Kosice-old, Košice
  - Detska fakultna nemocnica Kosice, Košice
  - Lipmet, s.r.o., Poprad
  - Fakultna nemocnica Trencin, Trenčín
- Spain (5):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Merida, Mérida, Badajoz
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
- Dr. med. Jean-Marc Nuoffer, Ch-3010 Bern, Switzerland
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty. Department of Pediatrics. Nutrition and Metabolism Unit, Ankara
  - Gazi University, Medical Faculty, Ankara
  - Ege University Medical Faculty, Izmir

REFERENCES:
- [Derived] Langslet G, Breazna A, Drogari E. A 3-year study of atorvastatin in children and adolescents with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2016 Sep-Oct;10(5):1153-1162.e3. doi: 10.1016/j.jacl.2016.05.010. Epub 2016 Jun 7. PMID 27678432
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581173&StudyName=Atorvastatin%20Three%20Year%20Pediatric%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin (5-80 mg): Tanner_Stage 1: Participants aged 6 to less than (<)10 years, at Tanner_Stage 1 received an initial dose of atorvastatin tablets, 5 milligrams per day (mg/day), orally (PO), through Week 4; after Week 4, dose may have been doubled to 10 mg/day, with subsequent doubling to 20 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target low-density lipoprotein cholesterol (LDL-C) (<3.35 millimoles per liter [mmol/L]) was not attained.
- Atorvastatin (10-80 mg): Tanner_Stage 2+: Participants aged greater than or equal to (≥) 10 to 15 years, at Tanner_Stage 2+ received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
Period: Overall Study
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Started | 139 | 132
Completed | 112 | 94
Not Completed | 27 | 38
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Pregnancy | 0 | 1
Not completed — Other | 5 | 13
Not completed — LDL below 2.59 mmol/L | 4 | 12
Not completed — Adverse Event | 4 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who took at least one dose of study drug.
Groups:
- Atorvastatin (5-80 mg): Tanner_Stage 1: Participants aged 6 to <10 years, at Tanner_Stage 1 received an initial dose of atorvastatin tablets, 5 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 10 mg/day, with subsequent doubling to 20 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
- Atorvastatin (10-80 mg): Tanner_Stage 2+: Participants aged ≥10 to 15 years, at Tanner_Stage 2+ received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
- Total: Total of all reporting groups
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+ | Total
Number analyzed (Participants) | 139 | 132 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.86) | 12.0 (1.68) | 10.2 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 79 | 125
  Male | 93 | 53 | 146

OUTCOME MEASURES:

1. Primary Outcome: Low Density Lipoprotein Cholesterol (LDL-C; Millimoles Per Liter [mMol/L]) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36 (or early termination [ET])
Population: FAS; n (number) equals (=) number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 139 | 132
mMol/L
  Baseline (n=139,132) | 6.304 (1.3130) | 5.921 (1.1646)
  Month 1 (n=131,130) | 4.087 (1.0264) | 3.675 (0.8749)
  Change at Month 1 (n=131,130) | -2.214 (0.7568) | -2.233 (0.8009)
  Month 2 (n=132,122) | 3.719 (0.8346) | 3.437 (0.7438)
  Change at Month 2 (n=132,122) | -2.586 (0.9297) | -2.554 (0.9155)
  Month 3 (n=126,117) | 3.503 (0.7566) | 3.270 (0.6533)
  Change at Month 3 (n=126,117) | -2.798 (1.0251) | -2.795 (1.0835)
  Month 6 (n=127,115) | 3.366 (0.5787) | 3.347 (0.5953)
  Change at Month 6 (n=127,115) | -2.968 (1.1096) | -2.732 (1.0660)
  Month 12 (n=121,109) | 3.409 (0.7395) | 3.196 (0.6565)
  Change at Month 12 (n=121,109) | -2.966 (1.0987) | -2.838 (1.1450)
  Month 18 (n=116,101) | 3.309 (0.5933) | 3.261 (0.5288)
  Change at Month 18 (n=116,101) | -3.105 (1.1558) | -2.835 (1.2128)
  Month 24 (n=111,96) | 3.316 (0.6803) | 3.189 (0.6537)
  Change at Month 24 (n=111,96) | -3.088 (1.2026) | -2.933 (1.2292)
  Month 30 (n=112,94) | 3.335 (0.6490) | 3.142 (0.6916)
  Change at Month 30 (n=112,94) | -3.090 (1.2402) | -3.008 (1.1489)
  Month 36/ET (n=123,117) | 3.450 (0.7372) | 3.457 (0.8808)
  Change at Month 36/ET (n=123,117) | -2.855 (1.2625) | -2.468 (1.3270)

2. Primary Outcome: Percent Change From Baseline in LDL-C
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36 (or ET)
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 132 | 130
percent change
  Month 1 (n=131,130) | -34.995 (9.7300) | -37.516 (10.0245)
  Month 2 (n=132,122) | -40.371 (9.6468) | -41.939 (10.4816)
  Month 3 (n=126,117) | -43.568 (10.2149) | -44.887 (12.7530)
  Month 6 (n=127,115) | -45.647 (9.6969) | -43.697 (11.1836)
  Month 12 (n=121,109) | -45.530 (10.5112) | -45.727 (13.5336)
  Month 18 (n=116,101) | -47.101 (10.5592) | -44.818 (13.2623)
  Month 24 (n=111,96) | -46.944 (11.9490) | -46.417 (13.8658)
  Month 30 (n=112,94) | -46.631 (12.0206) | -47.734 (12.6696)
  Month 36/ET (n=123,117) | -43.785 (13.5585) | -39.863 (17.5411)

3. Primary Outcome: High-Density Lipoprotein Cholesterol (HDL-C; mMol/L) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 139 | 132
mMol/L
  Baseline (n=139,132) | 1.349 (0.2732) | 1.277 (0.2546)
  Month 1 (n=131,130) | 1.360 (0.2717) | 1.292 (0.2650)
  Change at Month 1 (n=131,130) | 0.010 (0.1685) | 0.016 (0.1740)
  Month 2 (n=132,122) | 1.364 (0.2805) | 1.297 (0.2625)
  Change at Month 2 (n=132,122) | 0.014 (0.2238) | 0.025 (0.1600)
  Month 3 (n=126,117) | 1.371 (0.2768) | 1.274 (0.2606)
  Change at Month 3 (n=126,117) | 0.015 (0.1943) | 0.011 (0.1837)
  Month 6 (n=127,115) | 1.337 (0.2834) | 1.268 (0.2311)
  Change at Month 6 (n=127,115) | -0.011 (0.1848) | 0.010 (0.1833)
  Month 12 (n=121,109) | 1.328 (0.2885) | 1.241 (0.2429)
  Change at Month 12 (n=121,109) | -0.012 (0.1945) | -0.023 (0.1727)
  Month 18 (n=116,102) | 1.367 (0.3003) | 1.234 (0.2349)
  Change at Month 18 (n=116,102) | 0.024 (0.1923) | -0.027 (0.1744)
  Month 24 (n=111,96) | 1.385 (0.2729) | 1.266 (0.2443)
  Change at Month 24 (n=111,96) | 0.027 (0.2043) | 0.007 (0.1910)
  Month 30 (n=112,94) | 1.380 (0.2942) | 1.265 (0.2487)
  Change at Month 30 (n=112,94) | 0.032 (0.1997) | 0.006 (0.2150)
  Month 36/ET (n=123,117) | 1.335 (0.2918) | 1.278 (0.2516)
  Change at Month 36/ET (n=123,117) | -0.024 (0.1949) | 0.005 (0.1975)

4. Primary Outcome: Percent Change From Baseline in HDL-C
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 132 | 130
percent change
  Month 1 (n=131,130) | 1.526 (12.7845) | 2.192 (14.0769)
  Month 2 (n=132,122) | 2.195 (15.6882) | 2.544 (12.7802)
  Month 3 (n=126,117) | 1.929 (14.7329) | 1.674 (14.9525)
  Month 6 (n=127,115) | -0.016 (14.8853) | 1.877 (14.9113)
  Month 12 (n=121,109) | -0.069 (15.2821) | -1.023 (14.1983)
  Month 18 (n=116,102) | 2.472 (14.8939) | -1.165 (14.3783)
  Month 24 (n=111,96) | 3.014 (14.9559) | 1.737 (15.6924)
  Month 30 (n=112,94) | 3.345 (15.5080) | 1.868 (17.2633)
  Month 36/ET (n=123,117) | -1.125 (14.7816) | 1.602 (15.4895)

5. Primary Outcome: Total Cholesterol (mMol/L) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 139 | 132
mMol/L
  Baseline (n=139,132) | 8.056 (1.3356) | 7.647 (1.2250)
  Month 1 (n=134,131) | 5.785 (1.0497) | 5.352 (0.9345)
  Change at Month 1 (n=134,131) | -2.266 (0.7957) | -2.297 (0.8516)
  Month 2 (n=132,124) | 5.435 (0.8629) | 5.061 (0.7865)
  Change at Month 2 (n=132,124) | -2.620 (0.9581) | -2.654 (0.9707)
  Month 3 (n=127,118) | 5.195 (0.8000) | 4.883 (0.7034)
  Change at Month 3 (n=127,118) | -2.869 (1.0904) | -2.883 (1.1363)
  Month 6 (n=127,115) | 5.019 (0.6380) | 4.982 (0.6620)
  Change at Month 6 (n=127,115) | -3.063 (1.1687) | -2.809 (1.1133)
  Month 12 (n=121,109) | 5.081 (0.7470) | 4.799 (0.7176)
  Change at Month 12 (n=121,109) | -3.040 (1.1353) | -2.945 (1.2112)
  Month 18 (n=116,101) | 4.989 (0.6512) | 4.845 (0.5401)
  Change at Month 18 (n=116,101) | -3.168 (1.1990) | -2.965 (1.2667)
  Month 24 (n=111,96) | 5.032 (0.7111) | 4.817 (0.7413)
  Change at Month 24 (n=111,96) | -3.123 (1.2039) | -3.009 (1.2871)
  Month 30 (n=112,95) | 5.075 (0.6951) | 4.795 (0.8256)
  Change at Month 30 (n=112,95) | -3.096 (1.2999) | -3.048 (1.2716)
  Month 36/ET (n=123,117) | 5.134 (0.7863) | 5.099 (0.9318)
  Change at Month 36/ET (n=123,117) | -2.923 (1.3256) | -2.543 (1.3669)

6. Primary Outcome: Percent Change From Baseline in Total Cholesterol
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 134 | 131
percent change
  Month 1 (n=134,131) | -27.879 (8.2639) | -29.653 (8.5987)
  Month 2 (n=132,124) | -31.900 (8.5025) | -33.726 (9.2319)
  Month 3 (n=127,118) | -34.784 (9.4141) | -36.126 (11.0136)
  Month 6 (n=127,115) | -36.889 (9.2297) | -35.055 (10.0273)
  Month 12 (n=121,109) | -36.541 (9.2486) | -36.943 (11.9418)
  Month 18 (n=116,101) | -37.772 (9.7325) | -36.634 (11.4572)
  Month 24 (n=111,96) | -37.287 (9.9578) | -37.317 (12.2461)
  Month 30 (n=112,95) | -36.662 (11.2064) | -37.856 (12.5116)
  Month 36/ET (n=123,117) | -35.063 (12.0345) | -32.013 (14.5000)

7. Primary Outcome: Trigylcerides (mMol/L) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 139 | 132
mMol/L
  Baseline (n=139,132) | 0.880 (0.4343) | 0.980 (0.4986)
  Month 1 (n=134,131) | 0.759 (0.3958) | 0.815 (0.3848)
  Change at Month 1 (n=134,131) | -0.121 (0.3895) | -0.166 (0.5024)
  Month 2 (n=132,124) | 0.772 (0.3837) | 0.741 (0.3382)
  Change at Month 2 (n=132,124) | -0.103 (0.3652) | -0.246 (0.4825)
  Month 3 (n=127,118) | 0.699 (0.2916) | 0.748 (0.3357)
  Change at Month 3 (n=127,118) | -0.166 (0.3937) | -0.237 (0.4466)
  Month 6 (n=127,115) | 0.691 (0.3602) | 0.801 (0.3848)
  Change at Month 6 (n=127,115) | -0.183 (0.4305) | -0.188 (0.4880)
  Month 12 (n=121,109) | -0.747 (0.3901) | 0.789 (0.4050)
  Change at Month 12 (n=121,109) | -0.136 (0.4060) | -0.181 (0.5255)
  Month 18 (n=116,102) | 0.687 (0.3435) | 0.765 (0.3438)
  Change at Month 18 (n=116,102) | -0.190 (0.3665) | -0.219 (0.4623)
  Month 24 (n=111,96) | 0.725 (0.3676) | 0.790 (0.3651)
  Change at Month 24 (n=111,96) | -0.133 (0.4112) | -0.179 (0.4956)
  Month 30 (n=112,95) | 0.788 (0.3454) | 0.781 (0.4167)
  Change at Month 30 (n=112,95) | -0.082 (0.3898) | -0.187 (0.5728)
  Month 36/ET (n=123,117) | 0.764 (0.4220) | 0.794 (0.3894)
  Change at Month 36/ET (n=123,117) | -0.092 (0.4615) | -0.171 (0.5216)

8. Primary Outcome: Percent Change From Baseline in Trigylcerides
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 134 | 131
percent change
  Month 1 (n=134,131) | -5.950 (39.0995) | -5.927 (51.1811)
  Month 2 (n=132,124) | -3.260 (42.5136) | -14.832 (40.4952)
  Month 3 (n=127,118) | -8.760 (41.1184) | -14.415 (39.9951)
  Month 6 (n=127,115) | -11.817 (41.9879) | -9.097 (43.0350)
  Month 12 (n=121,109) | -7.981 (40.4511) | -7.950 (48.7238)
  Month 18 (n=116,102) | -13.113 (39.3990) | -12.443 (37.3822)
  Month 24 (n=111,96) | -6.697 (38.7027) | -7.328 (45.3694)
  Month 30 (n=112,95) | 0.657 (43.3886) | -4.935 (63.1887)
  Month 36/ET (n=123,117) | -0.703 (50.6333) | -7.759 (45.6372)

9. Primary Outcome: Very Low-Density Lipoprotein (VLDL; mMol/L) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 139 | 132
mMol/L
  Baseline (n=139,132) | 0.403 (0.1993) | 0.449 (0.2288)
  Month 1 (n=134,131) | 0.348 (0.1823) | 0.374 (0.1770)
  Change at Month 1 (n=134,131) | -0.056 (0.1793) | -0.076 (0.2307)
  Month 2 (n=132,124) | 0.354 (0.1757) | 0.340 (0.1541)
  Change at Month 2 (n=132,124) | -0.047 (0.1672) | -0.113 (0.2215)
  Month 3 (n=127,118) | 0.320 (0.1333) | 0.344 (0.1548)
  Change at Month 3 (n=127,118) | -0.076 (0.1805) | -0.108 (0.2044)
  Month 6 (n=127,115) | 0.317 (0.1652) | 0.367 (0.1767)
  Change at Month 6 (n=127,115) | -0.084 (0.1977) | -0.086 (0.2240)
  Month 12 (n=121,109) | 0.343 (0.1786) | 0.362 (0.1862)
  Change at Month 12 (n=121,109) | -0.062 (0.1872) | -0.082 (0.2421)
  Month 18 (n=116,101) | 0.315 (0.1571) | 0.349 (0.1571)
  Change at Month 18 (n=116,101) | -0.087 (0.1680) | -0.102 (0.2126)
  Month 24 (n=111,96) | 0.332 (0.1680) | 0.363 (0.1680)
  Change at Month 24 (n=111,96) | -0.061 (0.1887) | -0.081 (0.2285)
  Month 30 (n=112,95) | 0.361 (0.1581) | 0.358 (0.1914)
  Change at Month 30 (n=112,95) | -0.038 (0.1781) | -0.086 (0.2621)
  Month 36/ET (n=123,117) | 0.350 (0.1930) | 0.364 (0.1782)
  Change at Month 36/ET (n=123,117) | -0.042 (0.2112) | -0.079 (0.2385)

10. Primary Outcome: Percent Change From Baseline in VLDL
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 134 | 131
percent change
  Month 1 (n=134,131) | -6.060 (39.3300) | -5.805 (51.7264)
  Month 2 (n=132,124) | -3.097 (42.3626) | -14.694 (40.1710)
  Month 3 (n=127,118) | -8.711 (41.2631) | -14.263 (39.7239)
  Month 6 (n=127,115) | -11.591 (42.4219) | -9.158 (43.1397)
  Month 12 (n=121,109) | -7.739 (40.7579) | -7.827 (48.9819)
  Month 18 (n=116,101) | -12.911 (39.7908) | -12.768 (37.4142)
  Month 24 (n=111,96) | -6.654 (38.7945) | -6.920 (46.3317)
  Month 30 (n=112,95) | 0.627 (43.6239) | -4.751 (64.2502)
  Month 36/ET (n=123,117) | -0.520 (51.3422) | -7.842 (45.4640)

11. Primary Outcome: Apoliprotein A-1 (Apo A-1; Grams Per Liter [g/L]) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 138 | 132
g/L
  Baseline (n=138,132) | 1.396 (0.1839) | 1.308 (0.2006)
  Month 1 (n=132,130) | 1.419 (0.2233) | 1.337 (0.1927)
  Change at Month 1 (n=132,130) | 0.025 (0.1639) | 0.032 (0.1506)
  Month 2 (n=131,123) | 1.411 (0.1952) | 1.334 (0.1950)
  Change at Month 2 (n=131,123) | 0.016 (0.1519) | 0.025 (0.1355)
  Month 3 (n=126,117) | 1.405 (0.1914) | 1.306 (0.1919)
  Change at Month 3 (n=126,117) | 0.005 (0.1713) | 0.006 (0.1557)
  Month 6 (n=123,110) | 1.386 (0.2081) | 1.329 (0.1894)
  Change at Month 6 (n=123,110) | -0.007 (0.1609) | 0.026 (0.1818)
  Month 12 (n=120,108) | 1.347 (0.1893) | 1.271 (0.1798)
  Change at Month 12 (n=120,108) | -0.041 (0.1574) | -0.028 (0.1586)
  Month 18 (n=114,100) | 1.339 (0.1972) | 1.266 (0.1676)
  Change at Month 18 (n=114,100) | -0.049 (0.1558) | -0.038 (0.1643)
  Month 24 (n=113,95) | 1.364 (0.1929) | 1.275 (0.1736)
  Change at Month 24 (n=113,95) | -0.032 (0.1749) | -0.027 (0.1799)
  Month 30 (n=112,95) | 1.357 (0.2247) | 1.268 (0.1848)
  Change at Month 30 (n=112,95) | -0.040 (0.1857) | -0.036 (0.1861)
  Month 36/ET (n=125,118) | 1.327 (0.2081) | 1.272 (0.1664)
  Change at Month 36/ET (n=125,118) | -0.073 (0.1725) | -0.040 (0.1676)

12. Primary Outcome: Percent Change From Baseline in Apo A-1
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 132 | 130
percent change
  Month 1 (n=132,130) | 2.229 (12.4001) | 3.301 (12.2009)
  Month 2 (n=131,123) | 1.701 (11.0364) | 2.499 (10.7656)
  Month 3 (n=126,117) | 1.041 (12.4204) | 1.192 (12.1640)
  Month 6 (n=123,110) | -0.069 (12.1109) | 3.011 (14.1347)
  Month 12 (n=120,108) | -2.365 (11.5882) | -1.370 (12.3901)
  Month 18 (n=114,100) | -3.042 (11.2219) | -1.980 (12.2170)
  Month 24 (n=113,95) | -1.611 (12.4618) | -0.961 (13.9868)
  Month 30 (n=112,95) | -2.342 (13.3357) | -1.695 (14.2732)
  Month 36/ET (n=125,118) | -4.804 (12.0443) | -1.954 (12.7229)

13. Primary Outcome: Apoliprotein B (Apo B; g/L) During the Study
Description: Assessments were performed in the fasting state (minimum 10-hour fast). Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 138 | 132
g/L
  Baseline (n=138,132) | 1.454 (0.2890) | 1.381 (0.2619)
  Month 1 (n=132,130) | 1.062 (0.2423) | 0.967 (0.2257)
  Change at Month 1 (n=132,130) | -0.395 (0.1599) | -0.415 (0.1691)
  Month 2 (n=131,123) | 0.980 (0.1929) | 0.916 (0.1813)
  Change at Month 2 (n=131,123) | -0.471 (0.1825) | -0.484 (0.1858)
  Month 3 (n=126,117) | 0.930 (0.1836) | 0.890 (0.1707)
  Change at Month 3 (n=126,117) | -0.522 (0.2152) | -0.518 (0.2184)
  Month 6 (n=123,110) | 0.919 (0.1557) | 0.910 (0.1683)
  Change at Month 6 (n=123,110) | -0.535 (0.2092) | -0.503 (0.2086)
  Month 12 (n=120,108) | 0.918 (0.1816) | 0.871 (0.1493)
  Change at Month 12 (n=120,108) | -0.548 (0.2131) | -0.530 (0.2194)
  Month 18 (n=114,100) | 0.893 (0.1546) | 0.882 (0.1293)
  Change at Month 18 (n=114,100) | -0.578 (0.2343) | -0.533 (0.2463)
  Month 24 (n=113,95) | 0.918 (0.1719) | 0.884 (0.1575)
  Change at Month 24 (n=113,95) | -0.551 (0.2353) | -0.535 (0.2344)
  Month 30 (n=112,95) | 0.910 (0.1723) | 0.885 (0.1717)
  Change at Month 30 (n=112,95) | -0.560 (0.2664) | -0.533 (0.2467)
  Month 36/ET (n=125,118) | 0.926 (0.1860) | 0.924 (0.2173)
  Change at Month 36/ET (n=125,118) | -0.520 (0.2730) | -0.450 (0.2748)

14. Primary Outcome: Percent Change From Baseline in Apo B
Description: Assessments were performed in the fasting state (minimum 10-hour fast).
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 132 | 130
percent change
  Month 1 (n=132,130) | -26.933 (9.5550) | -29.851 (10.3544)
  Month 2 (n=131,123) | -31.867 (9.2821) | -33.959 (9.9478)
  Month 3 (n=126,117) | -35.163 (10.5680) | -35.849 (11.6832)
  Month 6 (n=123,110) | -35.900 (9.3398) | -34.740 (10.7982)
  Month 12 (n=120,108) | -36.624 (9.7413) | -36.842 (11.6106)
  Month 18 (n=114,100) | -38.158 (10.4084) | -36.211 (12.7805)
  Month 24 (n=113,95) | -36.426 (11.4333) | -36.677 (12.1824)
  Month 30 (n=112,95) | -36.668 (12.8783) | -36.453 (13.6888)
  Month 36/ET (n=125,118) | -34.507 (14.0740) | -31.362 (16.4770)

15. Primary Outcome: Number of Participants With Shift From Baseline in Tanner_Stage by Timepoint and Baseline Tanner_Stage
Description: Tanner_Stage was assessed based on 2 components by gender, pubic hair and breasts for females and pubic hair and genitalia for males. If these values of components were not same, then the Tanner_Stage had the higher value of 2 components for each gender by visit.
Time Frame: Baseline, Months 6, 12, 18, 24, 30, and 36/ET
Population: FAS; n=number of participants assessed for the specific parameter at a given visit.
Measure: Number; unit: participants
Groups:
- Atorvastatin (5-80 mg): Baseline Tanner_Stage 1: Participants aged 6 to <10 years, at Tanner_Stage 1 received an initial dose of atorvastatin tablets, 5 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 10 mg/day, PO, with subsequent doubling to 20 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
- Atorvastatin (10-80 mg): Baseline Tanner_Stage 2: Participants aged ≥10 to 15 years, at Tanner_Stage 2 received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
- Atorvastatin (10-80 mg): Baseline Tanner_Stage 3: Participants aged ≥10 to 15 years, at Tanner_Stage 3 received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, PO, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
- Atorvastatin (10-80 mg): Baseline Tanner_Stage 4: Participants aged ≥10 to 15 years, at Tanner_Stage 4 received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, PO, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
- Atorvastatin (10-80 mg): Baseline Tanner_Stage 5: Participants aged ≥10 to 15 years, at Tanner_Stage 5 received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, PO, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
Arm/Group | Atorvastatin (5-80 mg): Baseline Tanner_Stage 1 | Atorvastatin (10-80 mg): Baseline Tanner_Stage 2 | Atorvastatin (10-80 mg): Baseline Tanner_Stage 3 | Atorvastatin (10-80 mg): Baseline Tanner_Stage 4 | Atorvastatin (10-80 mg): Baseline Tanner_Stage 5
Number analyzed (Participants) | 127 | 52 | 25 | 31 | 18
participants
  Tanner_Stage 1, Month 6 (n=126,48,25,27,15) | 107 | 0 | 0 | 0 | 0
  Tanner_Stage 2 , Month 6 (n=126,48,25,27,15) | 14 | 34 | 0 | 0 | 0
  Tanner_Stage 3, Month 6 (n=126,48,25,27,15) | 5 | 10 | 14 | 0 | 0
  Tanner_Stage 4, Month 6 (n=126,48,25,27,15) | 0 | 4 | 11 | 25 | 1
  Tanner_Stage 5, Month 6 (n=126,48,25,27,15) | 0 | 0 | 0 | 2 | 14
  Tanner_Stage 1, Month 12 (n=121,43,23,26,15) | 85 | 0 | 0 | 0 | 0
  Tanner_Stage 2, Month 12 (n=121,43,23,26,15) | 25 | 17 | 0 | 0 | 0
  Tanner_Stage 3, Month 12 (n=121,43,23,26,15) | 10 | 21 | 11 | 0 | 0
  Tanner_Stage 4, Month 12 (n=121,43,23,26,15) | 1 | 5 | 10 | 22 | 1
  Tanner_Stage 5, Month 12 (n=121,43,23,26,15) | 0 | 0 | 2 | 4 | 14
  Tanner_Stage 1, Month 18 (n=115,41, 21,25,14) | 63 | 0 | 0 | 0 | 0
  Tanner_Stage 2, Month 18 (n=115,41, 21,25,14) | 31 | 15 | 0 | 0 | 0
  Tanner_Stage 3, Month 18 (n=115,41, 21,25,14) | 18 | 16 | 6 | 0 | 0
  Tanner_Stage 4, Month 18 (n=115,41, 21,25,14) | 3 | 9 | 11 | 18 | 1
  Tanner_Stage 5, Month 18 (n=115,41, 21,25,14) | 0 | 1 | 4 | 7 | 13
  Tanner_Stage 1, Month 24 (n=113,38,19,22,14) | 51 | 0 | 0 | 0 | 0
  Tanner_Stage 2, Month 24 (n=113,38,19,22,14) | 33 | 9 | 0 | 0 | 0
  Tanner_Stage 3, Month 24 (n=113,38,19,22,14) | 20 | 14 | 2 | 0 | 0
  Tanner_Stage 4, Month 24 (n=113,38,19,22,14) | 9 | 12 | 13 | 13 | 1
  Tanner_Stage 5, Month 24 (n=113,38,19,22,14) | 0 | 3 | 4 | 9 | 13
  Tanner_Stage 1, Month 30 (n=111,38,19,23,14) | 39 | 0 | 0 | 0 | 0
  Tanner_Stage 2, Month 30 (n=111,38,19,23,14) | 32 | 3 | 0 | 0 | 0
  Tanner_Stage 3, Month 30 (n=111,38,19,23,14) | 26 | 11 | 1 | 0 | 0
  Tanner_Stage 4, Month 30 (n=111,38,19,23,14) | 14 | 18 | 9 | 11 | 1
  Tanner_Stage 5, Month 30 (n=111,38,19,23,14) | 0 | 6 | 9 | 12 | 13
  Tanner_Stage 1, Month 36/ET (n=127,52,25,31,18) | 41 | 0 | 0 | 0 | 0
  Tanner_Stage 2, Month 36/ET (n=127,52,25,31,18) | 31 | 6 | 0 | 0 | 0
  Tanner_Stage 3, Month 36/ET (n=127,52,25,31,18) | 25 | 10 | 2 | 0 | 0
  Tanner_Stage 4, Month 36/ET (n=127,52,25,31,18) | 25 | 24 | 13 | 12 | 0
  Tanner_Stage 5, Month 36/ET (n=127,52,25,31,18) | 5 | 12 | 10 | 19 | 18

16. Primary Outcome: Height (Centimeters [cm]) During the Study: Males
Description: Investigator assessment of height changes during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; only male participants were included in the analysis. n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Atorvastatin (5-80 mg): Participants aged 6 to <10 years, at Tanner_Stage 1 received an initial dose of atorvastatin tablets, 5 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 10 mg/day, PO, with subsequent doubling to 20 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained. Participants aged ≥10 to 15 years, at Tanner_Stage 2+ received an initial dose of atorvastatin tablets, 10 mg/day, PO, through Week 4; after Week 4, dose may have been doubled to 20 mg/day, with subsequent doubling to 40 mg/day (as necessary; maximum dose was 80 mg/day), PO, if target LDL-C (<3.35 mmol/L) was not attained.
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 146
cm
  Baseline (n=146) | 144.36 (16.004)
  Month 1 (n=141) | 145.21 (16.114)
  Change at Month 1 (n=141) | 0.68 (0.964)
  Month 2 (n=138) | 145.93 (16.302)
  Change at Month 2 (n=138) | 1.27 (0.964)
  Month 3 (n=133) | 146.00 (16.139)
  Change at Month 3 (n=133) | 1.72 (1.172)
  Month 6 (n=129) | 147.17 (16.033)
  Change at Month 6 (n=129) | 3.24 (1.485)
  Month 12 (n=123) | 150.75 (16.321)
  Change at Month 12 (n=123) | 6.67 (2.385)
  Month 18 (n=119) | 153.26 (16.388)
  Change at Month 18 (n=119) | 9.31 (2.978)
  Month 24 (n=114) | 156.03 (16.001)
  Change at Month 24 (n=114) | 12.11 (3.630)
  Month 30 (n=114) | 158.78 (15.770)
  Change at Month 30 (n=114) | 14.86 (4.403)
  Month 36/ET (n=134) | 160.59 (15.602)
  Change at Month 36/ET (n=134) | 15.53 (6.801)

17. Primary Outcome: Percent Change From Baseline in Height: Males
Description: Investigator assessment of height changes during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 141
percent change
  Month 1 (n=141) | 0.47 (0.689)
  Month 2 (n=138) | 0.88 (0.652)
  Month 3 (n=133) | 1.19 (0.777)
  Month 6 (n=129) | 2.25 (0.987)
  Month 12 (n=123) | 4.66 (1.606)
  Month 18 (n=119) | 6.53 (2.021)
  Month 24 (n=114) | 8.53 (2.607)
  Month 30 (n=114) | 10.49 (3.260)
  Month 36/ET (n=134) | 10.97 (5.010)

18. Primary Outcome: Height (cm) During the Study: Females
Description: Investigator assessment of height changes during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: FAS; only female participants were included in the analysis. n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 125
cm
  Baseline (n=125) | 145.28 (14.108)
  Month 1 (n=124) | 146.06 (14.045)
  Change at Month 1 (n=124) | 0.71 (1.378)
  Month 2 (n=119) | 146.57 (13.919)
  Change at Month 2 (n=119) | 1.19 (1.700)
  Month 3 (n=115) | 146.81 (13.838)
  Change at Month 3 (n=115) | 1.68 (1.278)
  Month 6 (n=113) | 147.87 (13.619)
  Change at Month 6 (n=113) | 2.77 (1.720)
  Month 12 (n=107) | 150.84 (12.968)
  Change at Month 12 (n=107) | 5.50 (2.992)
  Month 18 (n=99) | 152.77 (12.648)
  Change at Month 18 (n=99) | 7.41 (4.043)
  Month 24 (n=95) | 154.79 (11.913)
  Change at Month 24 (n=95) | 9.61 (5.120)
  Month 30 (n=93) | 156.43 (11.288)
  Change at Month 30 (n=93) | 11.23 (6.118)
  Month 36/ET (n=121) | 156.52 (11.032)
  Change at Month 36/ET (n=121) | 11.23 (7.551)

19. Primary Outcome: Percent Change From Baseline in Height: Females
Description: Investigator assessment of height changes during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 124
percent change
  Month 1 (n=124) | 0.51 (1.004)
  Month 2 (n=119) | 0.84 (1.220)
  Month 3 (n=115) | 1.20 (0.925)
  Month 6 (n=113) | 1.98 (1.291)
  Month 12 (n=107) | 3.93 (2.262)
  Month 18 (n=99) | 5.30 (3.036)
  Month 24 (n=95) | 6.93 (3.933)
  Month 30 (n=93) | 8.13 (4.740)
  Month 36/ET (n=121) | 8.14 (5.789)

20. Primary Outcome: Weight (Kilograms [kg]) During the Study: Males
Description: Investigator assessment of weight changes during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 146
kg
  Baseline (n=146) | 40.79 (14.079)
  Month 1 (n=141) | 41.18 (14.287)
  Change at Month 1 (n=141) | 0.36 (1.203)
  Month 2 (n=138) | 41.83 (14.467)
  Change at Month 2 (n=138) | 0.80 (1.422)
  Month 3 (n=133) | 41.68 (14.266)
  Change at Month 3 (n=133) | 1.08 (1.907)
  Month 6 (n=129) | 42.47 (14.564)
  Change at Month 6 (n=129) | 2.00 (2.528)
  Month 12 (n=123) | 45.29 (15.526)
  Change at Month 12 (n=123) | 4.65 (3.822)
  Month 18 (n=119) | 47.53 (16.164)
  Change at Month 18 (n=119) | 7.02 (4.432)
  Month 24 (n=114) | 49.77 (16.401)
  Change at Month 24 (n=114) | 9.27 (5.079)
  Month 30 (n=114) | 52.12 (17.100)
  Change at Month 30 (n=114) | 11.61 (6.032)
  Month 36/ET (n=134) | 53.50 (16.787)
  Change at Month 36/ET (n=134) | 12.35 (6.771)

21. Primary Outcome: Percent Change From Baseline in Weight: Males
Description: Investigator assessment of weight changes during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 141
percent change
  Month 1 (n=141) | 0.94 (2.739)
  Month 2 (n=138) | 2.04 (3.262)
  Month 3 (n=133) | 2.73 (4.317)
  Month 6 (n=129) | 5.09 (5.559)
  Month 12 (n=123) | 11.85 (8.172)
  Month 18 (n=119) | 18.03 (9.629)
  Month 24 (n=114) | 24.28 (11.696)
  Month 30 (n=114) | 30.46 (14.058)
  Month 36/ET (n=134) | 32.54 (17.409)

22. Primary Outcome: Weight (kg) During the Study: Females
Description: Investigator assessment of weight changes during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 125
kg
  Baseline (n=125) | 42.14 (14.038)
  Month 1 (n=125) | 42.50 (14.007)
  Change at Month 1 (n=125) | 0.36 (0.924)
  Month 2 (n=120) | 42.86 (14.209)
  Change at Month 2 (n=120) | 0.67 (1.338)
  Month 3 (n=115) | 43.34 (14.753)
  Change at Month 3 (n=115) | 1.24 (1.819)
  Month 6 (n=113) | 44.26 (15.027)
  Change at Month 6 (n=113) | 2.10 (2.409)
  Month 12 (n=107) | 46.61 (15.158)
  Change at Month 12 (n=107) | 4.41 (3.317)
  Month 18 (n=99) | 48.32 (14.670)
  Change at Month 18 (n=99) | 6.24 (4.291)
  Month 24 (n=95) | 50.13 (14.731)
  Change at Month 24 (n=95) | 8.55 (5.038)
  Month 30 (n=93) | 51.73 (14.681)
  Change at Month 30 (n=93) | 10.02 (6.127)
  Month 36/ET (n=121) | 51.55 (14.498)
  Change at Month 36/ET (n=121) | 9.77 (7.047)

23. Primary Outcome: Percent Change From Baseline in Weight: Females
Description: Investigator assessment of weight changes during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 125
percent change
  Month 1 (n=125) | 0.97 (2.303)
  Month 2 (n=120) | 1.85 (3.206)
  Month 3 (n=115) | 3.16 (4.149)
  Month 6 (n=113) | 5.37 (5.529)
  Month 12 (n=107) | 11.65 (8.391)
  Month 18 (n=99) | 16.79 (11.315)
  Month 24 (n=95) | 23.43 (14.333)
  Month 30 (n=93) | 27.83 (17.507)
  Month 36/ET (n=121) | 27.26 (21.389)

24. Primary Outcome: Body Mass Index (BMI in kg Per Square Meter [kg/m^2]) During the Study: Males
Description: Investigator assessment of BMI changes during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 146
kg/m^2
  Baseline (n=146) | 18.97 (3.664)
  Month 1 (n=141) | 18.94 (3.751)
  Change at Month 1 (n=141) | 0.01 (0.577)
  Month 2 (n=138) | 19.06 (3.755)
  Change at Month 2 (n=138) | 0.06 (0.658)
  Month 3 (n=133) | 18.99 (3.745)
  Change at Month 3 (n=133) | 0.07 (0.890)
  Month 6 (n=129) | 19.04 (3.881)
  Change at Month 6 (n=129) | 0.10 (1.218)
  Month 12 (n=123) | 19.34 (3.922)
  Change at Month 12 (n=123) | 0.37 (1.541)
  Month 18 (n=119) | 19.65 (4.053)
  Change at Month 18 (n=119) | 0.73 (1.625)
  Month 24 (n=114) | 19.91 (4.098)
  Change at Month 24 (n=114) | 0.99 (1.745)
  Month 30 (n=114) | 20.18 (4.400)
  Change at Month 30 (n=114) | 1.25 (2.099)
  Month 36/ET (n=134) | 20.28 (4.137)
  Change at Month 36/ET (n=134) | 1.33 (1.958)

25. Primary Outcome: Percent Change From Baseline in BMI: Males
Description: Investigator assessment of BMI changes during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 141
percent change
  Month 1 (n=141) | 0.03 (2.953)
  Month 2 (n=138) | 0.31 (3.405)
  Month 3 (n=133) | 0.39 (4.496)
  Month 6 (n=129) | 0.55 (5.673)
  Month 12 (n=123) | 2.10 (7.065)
  Month 18 (n=119) | 3.98 (7.533)
  Month 24 (n=114) | 5.45 (8.306)
  Month 30 (n=114) | 6.80 (9.737)
  Month 36/ET (n=134) | 7.31 (9.290)

26. Primary Outcome: BMI (kg/m^2) During the Study: Females
Description: Investigator assessment of BMI changes during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 125
kg/m^2
  Baseline (n=125) | 19.44 (3.994)
  Month 1 (n=124) | 19.45 (3.973)
  Change at Month 1 (n=124) | -0.02 (0.582)
  Month 2 (n=119) | 19.47 (3.940)
  Change at Month 2 (n=119) | 0.00 (0.756)
  Month 3 (n=115) | 19.54 (4.171)
  Change at Month 3 (n=115) | 0.13 (0.861)
  Month 6 (n=113) | 19.68 (4.288)
  Change at Month 6 (n=113) | 0.24 (1.004)
  Month 12 (n=107) | 19.98 (4.257)
  Change at Month 12 (n=107) | 0.60 (1.305)
  Month 18 (n=99) | 20.24 (3.990)
  Change at Month 18 (n=99) | 0.92 (1.432)
  Month 24 (n=95) | 20.50 (3.976)
  Change at Month 24 (n=95) | 1.38 (1.624)
  Month 30 (n=93) | 20.75 (4.014)
  Change at Month 30 (n=93) | 1.59 (1.931)
  Month 36/ET (n=121) | 20.71 (4.217)
  Change at Month 36/ET (n=121) | 1.46 (1.948)

27. Primary Outcome: Percent Change From Baseline in BMI: Females
Description: Investigator assessment of BMI changes during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 124
percent change
  Month 1 (n=124) | -0.06 (3.058)
  Month 2 (n=119) | 0.16 (3.777)
  Month 3 (n=115) | 0.73 (4.314)
  Month 6 (n=113) | 1.26 (4.992)
  Month 12 (n=107) | 3.33 (6.765)
  Month 18 (n=99) | 5.14 (7.578)
  Month 24 (n=95) | 7.68 (8.661)
  Month 30 (n=93) | 8.89 (9.916)
  Month 36/ET (n=121) | 8.06 (10.147)

28. Primary Outcome: Age (Years) During the Study: Males
Description: Investigator assessment of age during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 146
years
  Baseline (n=146) | 9.94 (2.489)
  Month 1 (n=141) | 10.05 (2.553)
  Change at Month 1 (n=141) | 0.11 (0.309)
  Month 2 (n=138) | 10.14 (2.583)
  Change at Month 2 (n=138) | 0.18 (0.387)
  Month 3 (n=133) | 10.21 (2.567)
  Change at Month 3 (n=133) | 0.29 (0.457)
  Month 6 (n=129) | 10.43 (2.552)
  Change at Month 6 (n=129) | 0.55 (0.499)
  Month 12 (n=123) | 10.96 (2.543)
  Change at Month 12 (n=123) | 1.02 (0.155)
  Month 18 (n=119) | 11.47 (2.544)
  Change at Month 18 (n=119) | 1.54 (0.501)
  Month 24 (n=114) | 11.93 (2.534)
  Change at Month 24 (n=114) | 2.02 (0.132)
  Month 30 (n=114) | 12.46 (2.553)
  Change at Month 30 (n=114) | 2.54 (0.500)
  Month 36/ET (n=134) | 12.69 (2.587)
  Change at Month 36/ET (n=134) | 2.67 (0.899)

29. Primary Outcome: Percent Change From Baseline in Age: Males
Description: Investigator assessment of age during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 141
percent change
  Month 1 (n=141) | 1.09 (3.327)
  Month 2 (n=138) | 1.86 (4.184)
  Month 3 (n=133) | 3.16 (5.175)
  Month 6 (n=129) | 6.06 (5.956)
  Month 12 (n=123) | 11.13 (3.878)
  Month 18 (n=119) | 16.82 (7.732)
  Month 24 (n=114) | 21.92 (6.623)
  Month 30 (n=114) | 27.67 (9.855)
  Month 36/ET (n=134) | 28.90 (13.486)

30. Primary Outcome: Age (Years) During the Study: Females
Description: Investigator assessment of age during the study. Change from baseline was also determined.
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 125
years
  Baseline (n=125) | 10.55 (2.421)
  Month 1 (n=125) | 10.66 (2.436)
  Change at Month 1 (n=125) | 0.11 (0.317)
  Month 2 (n=120) | 10.78 (2.430)
  Change at Month 2 (n=120) | 0.20 (0.402)
  Month 3 (n=115) | 10.75 (2.449)
  Change at Month 3 (n=115) | 0.28 (0.450)
  Month 6 (n=113) | 10.99 (2.477)
  Change at Month 6 (n=113) | 0.52 (0.502)
  Month 12 (n=107) | 11.50 (2.416)
  Change at Month 12 (n=107) | 0.99 (0.097)
  Month 18 (n=99) | 12.02 (2.503)
  Change at Month 18 (n=99) | 1.52 (0.502)
  Month 24 (n=95) | 12.42 (2.482)
  Change at Month 24 (n=95) | 1.98 (0.144)
  Month 30 (n=93) | 12.99 (2.564)
  Change at Month 30 (n=93) | 2.52 (0.502)
  Month 36/ET (n=121) | 13.07 (2.547)
  Change at Month 36/ET (n=121) | 2.54 (0.940)

31. Primary Outcome: Percent Change From Baseline in Age: Females
Description: Investigator assessment of age during the study.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30 and 36/ET
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg)
Number analyzed (Participants) | 125
percent change
  Month 1 (n=125) | 1.10 (3.169)
  Month 2 (n=120) | 2.00 (4.128)
  Month 3 (n=115) | 2.74 (4.549)
  Month 6 (n=113) | 5.18 (5.221)
  Month 12 (n=107) | 10.00 (2.811)
  Month 18 (n=99) | 15.20 (6.006)
  Month 24 (n=95) | 20.08 (5.298)
  Month 30 (n=93) | 25.35 (7.415)
  Month 36/ET (n=121) | 25.73 (12.168)

32. Secondary Outcome: Percentage of Participants With Overall Expected Maturation and Development Consistent With Expectations as Assessed by the Investigator
Time Frame: Baseline, Months 1, 2, 3, 6, 12, 18, 24, 30 and 36 (or early termination)
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 139 | 132
percentage of participants
  Baseline (n=139,132) | 99.3 | 100.0
  Month 1 (n=118,113) | 100.0 | 100.0
  Month 2 (n=116,109) | 100.0 | 100.0
  Month 3 (n=130,118) | 100.0 | 100.0
  Month 6 (n=127,115) | 100.0 | 99.1
  Month 12 (n=121,109) | 100.0 | 99.1
  Month 18 (n=115,102) | 100.0 | 100.0
  Month 24 (n=113,95) | 100.0 | 100.0
  Month 30 (n=111,94) | 100.0 | 98.9
  Month 36/Early Termination (n=128,127) | 99.2 | 99.2

33. Primary Outcome: Flow-Mediated Dilatation (FMD) During the Study
Description: Percent (%) FMD was calculated as (hyperemic diameter minus resting diameter) divided by the resting diameter multiplied by 100. Change from baseline was also determined.
Time Frame: Baseline, Months 6, 12, 18, 24, 30 and 36/ET
Population: FMD Set: all participants enrolled in the FMD study who had at least baseline FMD measurements. n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: % FMD
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 37 | 36
% FMD
  Baseline (n=37,36) | 5.523 (3.2062) | 6.651 (4.4926)
  Month 6 (n=27,23) | 5.749 (2.5047) | 6.520 (4.0763)
  Change at Month 6 (n=27,23) | -0.063 (3.4768) | -0.759 (4.8732)
  Month 12 (n=32,29) | 4.732 (1.8477) | 6.363 (8.0370)
  Change at Month 12 (n=32,29) | -0.952 (3.6796) | -0.778 (9.4743)
  Month 18 (n=33,28) | 4.942 (2.6740) | 4.668 (3.8874)
  Change at Month 18 (n=33,28) | -0.762 (3.7374) | -2.556 (6.3123)
  Month 24 (n=33,28) | 4.538 (2.4239) | 5.679 (4.3224)
  Change at Month 24 (n=33,28) | -1.166 (3.2524) | -1.545 (7.2325)
  Month 30 (n=33,28) | 5.571 (2.7198) | 5.191 (2.5120)
  Change at Month 30 (n=33,28) | -0.134 (3.3399) | -2.033 (5.8591)
  Month 36/ET (n=34,33) | 4.987 (2.2540) | 5.360 (2.9873)
  Change at Month 36/ET (n=34,33) | -0.550 (3.6625) | -1.563 (4.8355)

34. Primary Outcome: Percent Change From Baseline in FMD
Description: Percent (%) FMD was calculated as (hyperemic diameter minus resting diameter) divided by the resting diameter multiplied by 100.
Time Frame: Months 6, 12, 18, 24, 30 and 36/ET
Population: FMD Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 34 | 33
percent change
  Month 6 (n=27,23) | 14.867 (67.6028) | -0.205 (60.7192)
  Month 12 (n=32,29) | -3.880 (56.1910) | 15.444 (207.6932)
  Month 18 (n=33,28) | -4.598 (68.0267) | -24.387 (81.5683)
  Month 24 (n=33,28) | -9.992 (57.3868) | 3.850 (102.2001)
  Month 30 (n=33,28) | 7.000 (63.0894) | -18.804 (42.2259)
  Month 36/ET (n=34,33) | 0.648 (62.5814) | -7.506 (61.2361)

35. Secondary Outcome: Percentage of Participants by Study Drug Compliance Category
Description: Compliance to study drug was categorized as <80%, 80% - 120%, and greater than (>) 120%.
Time Frame: Months 1, 2, 3, 6, 12, 18, 24, 30, and 36 (or early termination)
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Number analyzed (Participants) | 135 | 132
percentage of participants
  Month 1, <80% (n=135,132) | 3.0 | 6.8
  Month 1, 80%-120% (n=135,132) | 97.0 | 93.2
  Month 1, >120% (n=135,132) | 0 | 0
  Month 2, <80% (n=132,126) | 6.8 | 7.9
  Month 2, 80%-120% (n=132,126) | 92.4 | 92.1
  Month 2, >120% (n=132,126) | 0.8 | 0
  Month 3, <80% (n=130,118) | 3.8 | 7.6
  Month 3, 80%-120% (n=130,118) | 95.4 | 92.4
  Month 3, >120% (n=130,118) | 0.8 | 0
  Month 6, <80% (n=127,115) | 7.9 | 9.6
  Month 6, 80%-120% (n=127,115) | 92.1 | 90.4
  Month 6, >120% (n=127,115) | 0 | 0
  Month 12, <80% (n=121,109) | 7.4 | 7.3
  Month 12, 80%-120% (n=121,109) | 92.6 | 92.7
  Month 12, >120% (n=121,109) | 0 | 0
  Month 18, <80% (n=116,102) | 4.3 | 5.9
  Month 18, 80%-120% (n=116,102) | 94.0 | 94.1
  Month 18, >120% (n=116,102) | 1.7 | 0
  Month 24, <80% (n=113,95) | 8.8 | 9.5
  Month 24, 80%-120% (n=113,95) | 91.2 | 89.5
  Month 24, >120% (n=113,95) | 0 | 1.1
  Month 30, <80% (n=112,94) | 8.0 | 6.4
  Month 30, 80%-120% (n=112,94) | 92.0 | 92.6
  Month 30, >120% (n=112,94) | 0 | 1.1
  Month 36/ET, <80% (n=129,129) | 11.6 | 16.3
  Month 36/ET, 80%-120% (n=129,129) | 86.8 | 83.7
  Month 36/ET, >120% (n=129,129) | 1.6 | 0

ADVERSE EVENTS:
Time Frame: Baseline up through Month 36
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Atorvastatin (5-80 mg): Tanner_Stage 1 | Atorvastatin (10-80 mg): Tanner_Stage 2+
Serious Adverse Events (participants affected / at risk) | 14/139 | 7/132
Other Adverse Events (participants affected / at risk) | 93/139 | 86/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (5-80 mg): Tanner_Stage 1 (N=139) | Atorvastatin (10-80 mg): Tanner_Stage 2+ (N=132)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Appendix disorder (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type I diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intravascular papillary endothelial hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Testsicular appendage torsion (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (5-80 mg): Tanner_Stage 1 (N=139) | Atorvastatin (10-80 mg): Tanner_Stage 2+ (N=132)
Abdominal pain (Gastrointestinal disorders) | 21 | 10
Nasopharyngitis (Infections and infestations) | 26 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 10
Headache (Nervous system disorders) | 25 | 25
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 3 | 8
Vomiting (Gastrointestinal disorders) | 15 | 7
Pyrexia (General disorders) | 15 | 13
Bronchitis (Infections and infestations) | 9 | 1
Ear infection (Infections and infestations) | 9 | 6
Gastroenteritis (Infections and infestations) | 17 | 12
Influenza (Infections and infestations) | 13 | 14
Pharyngitis (Infections and infestations) | 9 | 8
Respiratory tract infection (Infections and infestations) | 7 | 0
Rhinitis (Infections and infestations) | 13 | 9
Tonsillitis (Infections and infestations) | 10 | 6
Upper respiratory tract infection (Infections and infestations) | 20 | 10
Viral upper respiratory tract infection (Infections and infestations) | 13 | 3
Blood creatine phosphokinase increased (Investigations) | 3 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.